CLINICAL TRIAL: NCT06909669
Title: Ultra-brief Psychological Treatments for Emocional Symptoms and Disorders: An Efficacy and Efficiency Analysis
Brief Title: Ultra-brief Psychological Treatments for Emotional Symptoms and Disorders
Acronym: UltraPsyBrief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: State Research Agency, Spain (Other Government); University Hospital Reina Sofia, Cordoba (Unknown)
Responsible Party: Principal Investigator, Juan A. Moriana, Professor, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2023-152589OB-I00
Record Dates: First submitted 2025-03-07; First posted 2025-04-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder; Generalized Anxiety Disorder; Generalized Anxiety; Anxiety; Somatoform Disorders; Somatic Symptom Disorder (DSM-5); Somatization; Emotional Disorders
Keywords: ultra-brief therapy; brief therapy; transdiagnostic therapy; cognitive-behavioral therapy; randomized controled trial
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders; Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial with pre-post measures and follow-ups.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Group brief TD-CBT (Experimental)
  Interventions: Behavioral: Group brief transdiagnostic cognitive-behavioral therapy
- Group 2: Group ultra-brief TD-CBT (Experimental)
  Interventions: Behavioral: Group ultra-brief transdiagnostic cognitive-behavioral therapy
- Group 3: Individual ultra-brief TD-CBT (Experimental)
  Interventions: Behavioral: Individual ultra-brief transdiagnostic cognitive-behavioral treatment format
- Group 4: relaxation (Active Comparator)
  Interventions: Behavioral: Group relaxation

INTERVENTIONS:
Behavioral: Group brief transdiagnostic cognitive-behavioral therapy — Eight-session treatment based on Barlow's Unified Protocol. These sessions include: improving motivation and commitment to treatment, understanding the functioning of emotions, emotional awareness training, developing more flexible and adaptive thinking patterns, reduction of emotional avoidance and emotion-driven behaviors; awareness and tolerance of physical sensations; interoceptive and situational emotional exposure; achievement, maintenance and relapse prevention. In addition, the intervention incorporates modules on behavioral activation and problem-solving.
  Arms: Group 1: Group brief TD-CBT
Behavioral: Group relaxation — The participants in this group will receive basic training in Jacobson's progressive relaxation with a similar periodicity to the ultra-brief intervention.
  Arms: Group 4: relaxation
Behavioral: Group ultra-brief transdiagnostic cognitive-behavioral therapy — This intervention consists of a four-session version of the brief transdiagnostic treatment (Experimental group 1). The reduced format preserves the principal treatment modules, including psychoeducation, emotion regulation, behavioral activation, and problem-solving.The reduction is achieved by combining sessions 1 and 2, eliminating 3 and 6 and combining sessions 7 and 8. Treatment groups will consist of 8-10 people. Each session will have a duration of 1.5 hours and the intervention will be carried out on a weekly basis, with a maximum duration of four weeks.
  Arms: Group 2: Group ultra-brief TD-CBT
Behavioral: Individual ultra-brief transdiagnostic cognitive-behavioral treatment format — Participants of this group, wil receive the same treatment than group 2 (ultra-brief transdiagnostic cognitive-behavioraltreatment in group format) but individual format. Each session will have a duration of 1 hour and the intervention will be carried out on a weekly basis, with a maximum duration of four weeks.
  Arms: Group 3: Individual ultra-brief TD-CBT

SUMMARY:
The main objective of this randomized clinical trial is to study if various modalities of brief (eight sessions) and ultra-brief (four sessions) transdiagnostic cognitive-behavioral treatment work for decrease emotional symptoms and disorders, as well as to find out which variables of cognition and of the intervention process itself are involved in the therapeutic improvement.

The investigators will compare the interventions of four groups: brief group treatment (1), ultra-brief group treatment (2), ultra-brief individual treatment (3) with the ultra-brief relaxation (control) group.

The main questions the study aims to answer are:

* Will the brief and ultra-brief treatment formats works better than the relaxation-based control group?
* Will results obtained between the brief group therapy group and the ultra-brief group therapy group be similar?
* Will the individual ultra brief therapy be more effective than the two group therapies because of common factors, such as the therapeutic alliance?
* Will group therapies be more beneficial for cost and in terms of capability to reduce emocional symptoms than individual therapy? Participants will be randomly assigned to each of the groups and will receive the corresponding treatment, with different number of sessions. They will answer a series of questionnaires at the beginning and at the end of the intervention, as well as 3 months and 6 months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients presenting negative emotional symptomatology (anxiety, depression or somatizations), mild or moderate. Specifically, they will be included in the study if they present a score ≥ 5 on the PHQ-9, the GAD-7 or the PHQ-15.

Exclusion Criteria:

* Bipolar disorder, personality disorder, psychosis or substance abuse, indicated by SCID-5-CV
* Recent suicide attempt.
* Severe emotional symptoms (PHQ-15 or GAD-7 ≥ 15; or PHQ-9 ≥ 20).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  The PHQ-9 is the depression module of the PHQ, that scores the 9 DSM-IV depression criteria present in the last two weeks from 0 ("not at all") to 3 ("nearly every day"). A score of 10 is usually set as the cut-off point for major depression disorder (MDD): a score of 10-14 indicates minor depression, moderate MDD, or dysthymia; 15-19, moderately severe MDD; and 20-27, severe MDD. This tool has been tested in Spanish primary care centres (McDonald's ω = .89).
Generalized Anxiety Disorder Scale (GAD-7) | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  The GAD-7 assesses common anxiety symptoms in the last two weeks, scoring from 0 ("not at all") to 3 ("nearly every day"). Cut points of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively. The algorithm sets 8 as the cut point for GAD, however it has been found that a score of 10 is more optimal. We will use a version validated in Spanish, that was recently tested in primary care centres (Cronbach's α = .83).
Patient Health Questionnaire-15 (PHQ-15) | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  The PHQ-15 is the somatization module of the PHQ. It includes 13 somatic symptoms plus 2 from the PHQ-9 (sleeping problems and fatigue). Scores of 5, 10, and 15 represent low, medium, and high somatic symptom severity, respectively. To screen a somatization disorder, whereas the original algorithm needs of at least a score of 2 in three or more somatic symptoms (sensitivity of 78% and specificity of 71%), the cut point usually used is 10; nevertheless, since this can be obtained with ten symptoms of mild severity, we decided to join both criteria to screen the disorder. Furthermore, an absence of biological cause is also often required (since PHQ-15 does not distinguish between medically explained and unexplained symptoms), but the self-administered nature of the PHQ-15 makes difficult to determine this. The PHQ-15 has been validated with Spanish psychiatric outpatients (α = .78).
Structured Clinical Interview for DSM-5, Clinical Version (SCID-5-CV) | Baseline and post-treatment (two weeks after the end of treatment).
  Structured Clinical Interview for DSM-5, Clinical Version (SCID-5-CV), is an interview commonly used to diagnose mental disorders according to the DSM-5 criteria. It is administered by a clinician or trained mental heatlh professional who is familiar with the DSM-5 classification and diagnostic criteria. We will use only the diagnostic criteria to evaluate the existence or not of Major Depressive Episode, Generalized Anxiety Disorder and to exclude the existence of other disorders such as Bipolar Disorder, psychotic disorders, substance use and personality disorder.

SECONDARY OUTCOMES:
Cognitive Emotional Regulation Questionnaire (CERQ-27) | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  It is a 27-item instrument (3 items for each subscale) that measures the following cognitive strategies of emotional regulation: self-blame, acceptance, rumination, refocusing on planning, positive reappraisal, putting into perspective, catastrophizing, and blaming others. Its psychometric properties are adequate, with a Cronbarch's α for each subscale between 0.73 and 0.88.
Common Factor Scale (MPOQ) | Peritreatment: weeks 1 and 3 (for 4-session groups); weeks 1 and 7 (for the 8-session group).
  This 14-item scale measures six different domains of common factors: task agreement, goal agreement, therapist empathy, therapist experience, treatment credibility, and expectations. The items are scored from 1 (strongly disagree) to 7 (strongly agree). This scale has two underlying factors, "Confidence in the therapist" and "Confidence in the treatment", which show an excellent internal consistency (α=.924 and α=.828, respectively).
Working Alliance Inventory-Short Form Patient version (WAI-S-P) | Peritreatment: weeks 1 and 3 (for 4-session groups); weeks 1 and 7 (for the 8-session group).
  We use the Bonding subscale from Working Alliance Inventory-Short Form Patient version. It consists of four items with 7 response options that score from 1 (never) to 7 (always). This scale has an excellent internal consistency (α=.93).
Psychological Outcome Profiles (PSYCHLOPS) | Baseline and post-treatment (two weeks after the end of treatment).
  Psychological Outcome Profiles is a individualized patiet-reported outcome measure that measures psychological distress. It includes four items covering three domains: (1) Problems (two free-text patient-generated items regarding the two problems that trouble him/her most, questions Q1 and Q2); (2) Function (one free-text patient-generated item corresponding to what has become hardest to do because of his/her problem(s), question Q3); and (3) Well-being (pre-set standardized item about how the patient felt in him/herself in the previous week, question Q4). Items are scored for intensity on a 6-point rating scale (from "Not affected at all" to "Severely affected") and for duration (from "Under 1 month" to "Over 5 years"). PSYCHLOPS total scoring is obtained by summing the scores of the four severity scales (Q1b, Q2b, Q3b, and Q4). PSYCHLOPS has good internal consistency (α = 0.82).
Satisfaction with therapy | Post-treatment (two weeks after the end of treatment).
  Satisfaction with therapy is a scale that collects different questions about the patient's subjective perception of therapy, including a question about expectations, difficulties during therapy and level of satisfaction. Some questions are formulated with an open response where they can describe and others with items ranging from 0 ("not at all") to 5 ("totally").
Sociodemographic data | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  Sociodemographic data includes information about gender, age, marital status, level of education, employment situation and level of income (per year)
Healthcare use questions | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  Questions on Health Care to find out about labor and health costs, addressing different issues such as visits made to health areas for own problems, medical tests, medications or other substances for anxiety and depression and/or to sleep better, in the last 30 days, and attendance to other psychological/psychiatric therapy, public or private different from the one offered.
Acceptance and Action Questionnaire (AAQ-II) | Baseline, post-treatment (two weeks after the end of treatment), and follow-ups (3 and 6 months)
  We used the Spanish adaptation. It is a 7-item instrument that measures psychological inflexibility or experiential avoidance. It is a self-report with 7 Likert-type items with 7 response options, where 1 means "never true" and 7 means "always true". A higher AAQ-II score suggests more psychological inflexibility. The scale measures the tendency to shy away from disagreeable experiences as well as a lack of contact with the present moment due to distress. The AAQ-II exhibited excellent consistency (α = 0.93).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Moriana Elvira Professor, Principal Investigator — Universidad de Córdoba
Locations (2):
- Spain (2):
  - Unidad de Salud Mental del Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Unidad de Atención Psicológica (UNAP) de la Universidad de Córdoba, Córdoba, Córdoba

REFERENCES:
- [Background] Ruiz, F. J., Suárez-Falcón, J. C., Cárdenas-Sierra, S., Durán, Y., Guerrero, K., & Riaño-Hernández, D. (2016). Psychometric properties of the Acceptance and Action Questionnaire-II in Colombia. The Psychological Record, 66, 429-437. https://doi.org/10.1007/s40732-016-0183-2
- [Result] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Result] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Result] Ros Montalban S, Comas Vives A, Garcia-Garcia M. Validation of the Spanish version of the PHQ-15 questionnaire for the evaluation of physical symptoms in patients with depression and/or anxiety disorders: DEPRE-SOMA study. Actas Esp Psiquiatr. 2010 Nov-Dec;38(6):345-57. Epub 2010 Nov 1. PMID 21188674
- [Result] Munoz-Navarro R, Cano-Vindel A, Moriana JA, Medrano LA, Ruiz-Rodriguez P, Aguero-Gento L, Rodriguez-Enriquez M, Piza MR, Ramirez-Manent JI. Screening for generalized anxiety disorder in Spanish primary care centers with the GAD-7. Psychiatry Res. 2017 Oct;256:312-317. doi: 10.1016/j.psychres.2017.06.023. Epub 2017 Jun 12. PMID 28666201
- [Result] Munoz-Navarro R, Cano-Vindel A, Medrano LA, Schmitz F, Ruiz-Rodriguez P, Abellan-Maeso C, Font-Payeras MA, Hermosilla-Pasamar AM. Utility of the PHQ-9 to identify major depressive disorder in adult patients in Spanish primary care centres. BMC Psychiatry. 2017 Aug 9;17(1):291. doi: 10.1186/s12888-017-1450-8. PMID 28793892
- [Result] Holgado-Tello, F., Amor, P.J., Lasa, A., & Domínguez, J. (2018). Two new brief versions of the cognitive emotion regulation questionnaire and its relationships with depression and anxiety. Anales de Psicología, 34(3), 458-464. https://doi.org/10.6018/analesps.34.3.306531
- [Result] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Result] First, M.B., Williams, J.B.W., Kats, R.S., Spitzer, R.(2016). Structured Clinical Interview for DSM-S Disorders-Clinician version (SCID-S-CV). Arlington, VA, American Psychiatric Association,
- [Result] Finsrud I, Nissen-Lie HA, Vrabel K, Hostmaelingen A, Wampold BE, Ulvenes PG. It's the therapist and the treatment: The structure of common therapeutic relationship factors. Psychother Res. 2022 Feb;32(2):139-150. doi: 10.1080/10503307.2021.1916640. Epub 2021 May 2. PMID 33938407
- [Result] Diez-Quevedo C, Rangil T, Sanchez-Planell L, Kroenke K, Spitzer RL. Validation and utility of the patient health questionnaire in diagnosing mental disorders in 1003 general hospital Spanish inpatients. Psychosom Med. 2001 Jul-Aug;63(4):679-86. doi: 10.1097/00006842-200107000-00021. PMID 11485122
- [Result] Ashworth, M., Shepherd, M., Christey, J., Matthews, V., Wright, K., Parmentier, H., Robinson, S., & Godfrey, E. (2004). A client-generated psychometric instrument: the development of 'PSYCHLOPS'. Counselling and Psychotherapy Research, 4, 27-31. https://doi.org/10.1080/14733140412331383913
- [Result] Andrade-González, N., y Fernández-Liria, A. (2016). Spanish adaptation of the Working Alliance Inventory-Short (WAI-S). Current Psychology: A Journal for Diverse Perspectives on Diverse Psychological Issues, 35(1), 169-177. https://doi.org/10.1007/s12144-015-9365-3